CLINICAL TRIAL: NCT00003045
Title: A Phase II Trial of Hyperthermia and Radiotherapy for Locally Advanced Adenocarcinoma of the Prostate
Brief Title: Hyperthermia Plus Radiation Therapy in Treating Patients With Nonmetastatic Advanced Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Irving Kaplan, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94-153; P30CA006516 (NIH); NCI-H97-1294
Record Dates: First submitted 1999-11-01; First posted 2003-07-11 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diathermy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hyperthermia (Experimental): XRT and Hyperthermia Post-therapy evaluation PSA, Clinical Exam, and Prostate Biopsy ( @ 12 Months)
  Interventions: Device: Hyperthermia; Radiation: XRT

INTERVENTIONS:
Device: Hyperthermia — Hyperthermia is delivered by the transrectal ultrasound applicator just prior to XRT, at least one week apart, during the first 4 weeks of XRT. The goal of hyperthermia is CEM T 90 43 greater than or equal to 10 minutes. The maximum applied power duration will be 120 minutes per treatment session
Radiation: XRT — external beam radiation to a dose of 4500 cGy to a small pelvic field, followed by a boost to a reduced volume for an additional 2160 cGy. XRT is given daily, 5 days a week for 180 cGy per day. Total radiation dose=6660cGy
  Other Names: Radiation Therapy

SUMMARY:
Hyperthermia therapy may kill prostate cancer cells by heating them to several degrees above body temperature. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining hyperthermia with radiation therapy may kill more tumor cells.

The purpose of this study is to determine the ability of hyperthermia when combined with radiation therapy and in some patients hormonal therapy to control prostate cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine the ability of hyperthermia (heat treatments produced by sound waves) when combined with radiation therapy and in some patients hormonal therapy to control prostate cancer.

Hyperthermia refers to the use of temperatures 42 oC (107-6oF) or higher to treatment malignant tumors. Laboratory and some clinical reports have demonstrated a tumor killing effect if tumors are heated to 43oC (109oF) for 30-60 minutes.

Many studies have shown that hyperthermia improves the killing effect of radiation treatments for many tumors. In clinical studies, the addition of hyperthermia has shown to be beneficial for tumors of the breast, urinary bladder and the head and neck region with combined with radiation therapy. Investigators found an improvement in tumor response rates and a lengthened duration of response. The proposed study is one of the first controlled studies to attempt to prove the usefulness of hyperthermia for patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria

* Histologic confirmation of prostate cancer. (Slides will be obtained for central review)
* Clinical stage T2b, T2c, T3a, or T3b disease as defined by the AJCC 4th edition staging manual (see Appendix A)
* No evidence of metastatic disease (bone, lymph node or visceral) based on bone scan and computed tomography
* Adequate hematologic function

  * WBC> 4000/mm3
  * platelet count > 100, 000/mm3
  * hematocrit of > 30%
* An ECOG Performance Status of zero or one
* Age ≥ 18
* A life expectancy of 5 years or more(excluding possible prostate related causes)

Exclusion Criteria :

* Prior history of malignancy (except for non-melanoma skin cancer)
* Prior systemic therapy

  * No prior chemotherapy
  * No prior hormonal therapy other than that recommended in this protocol
* Prior pelvic radiotherapy
* Medical problems (such as an abnormal bleeding propensity) which would make transrectal ultrasound-directed transperineal thermal probe placement hazardous.
* Patients with severe insulin-dependent diabetes mellitus and evidence of neuropathy or vaculopathy
* Patients with unstable cardiac status including:

  * Unstable angina pectoris on medication
  * Patients with documented myocardial infarction within six months of protocol entry
  * Congestive heart failure requiring medication
  * Patients on anti-arrhythmic drugs
  * Severe hypertension (diastolic BP> 100 on medication
  * Patients with cardiac pacemakers
* Severe cerebrovascular disease (multiple CVA or CVA within 6 months)
* Severe COPD (medication requiring, with FEV 1 < 50% of expected or < 1 liter)
* Individuals who appear unlikely to tolerate the required prolonged stationary position during treatment due to emotional immaturity or instability or otherwise due to mental incompetence.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1997-04; Primary Completion 2001-12-31 (Actual); Study Completion 2003-12-31 (Actual)

PRIMARY OUTCOMES:
Time of PSA Failure | 2 Years
  Kaplan Meier estimation and Cox regression model

SECONDARY OUTCOMES:
Local Control and Disease Specific survival | One year post treatment
  Local Control and Disease Specific survival

CONTACTS AND LOCATIONS:
Overall Officials: Irving Kaplan, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hurwitz MD, Kaplan ID, Hansen JL, Prokopios-Davos S, Topulos GP, Wishnow K, Manola J, Bornstein BA, Hynynen K. Association of rectal toxicity with thermal dose parameters in treatment of locally advanced prostate cancer with radiation and hyperthermia. Int J Radiat Oncol Biol Phys. 2002 Jul 15;53(4):913-8. doi: 10.1016/s0360-3016(02)02809-2. PMID 12095557
- [Background] Hurwitz MD, Kaplan ID, Svensson GK, Hynynen K, Hansen MS. Feasibility and patient tolerance of a novel transrectal ultrasound hyperthermia system for treatment of prostate cancer. Int J Hyperthermia. 2001 Jan-Feb;17(1):31-7. doi: 10.1080/02656730150201570. PMID 11212878